CLINICAL TRIAL: NCT01950793
Title: Steroid Versus Hyaluronic Acid Ultrasound-guided Injection for Trigger Finger: A Comparative Study of Outcomes
Brief Title: A Comparison Between Sonoguided Injection Corticosteroid and Hyaluronic Acid Injection in Treatment of Trigger Finger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-11-001A
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Trigger Finger
Keywords: Hyaluronic acid, trigger finger
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Triamcinolone Acetonide; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- steroid (Active Comparator): used ultrasound-guided inject 1c.c triamcinolone acetonide 10mg/mL (Shincort®, YSP, Taiwan)into the sheath of the flexor tendons, penetrated to the A1 pulley.
  One injection only
  Interventions: Drug: triamcinolone acetonide
- Hyaluronic acid (Experimental): used ultrasound-guided inject 1c.c Hyaluronic acid (Artz®, Seikagaku, Japan)into the sheath of the flexor tendons, penetrated to the A1 pulley.
  One injection only
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Drug: triamcinolone acetonide — used ultrasound-guided inject 1c.c triamcinolone acetonide 10mg/mL (Shincort®, YSP, Taiwan)into the sheath of the flexor tendons, penetrated to the A1 pulley.
  One injection only Steroid
  Other Names: triamcinolone acetonide 10mg/mL (Shincort®, YSP, Taiwan)
  Arms: steroid
Drug: Hyaluronic Acid — used ultrasound-guided inject 1c.c Hyaluronic acid (Artz®, Seikagaku, Japan)into the sheath of the flexor tendons, penetrated to the A1 pulley.
  One injection only
  Other Names: Hyaluronic acid (Artz®, Seikagaku, Japan)
  Arms: Hyaluronic acid

SUMMARY:
The study is to compare the effect between steroid injection and Hyaluronic acid in treatment trigger finger. Using sonoguided injection technique achieves more accurate injection location and therapeutic effect. We hypothesize hyaluronic acid has both lubricant and anti-inflammation effect in treatment of trigger finger, and can provide better outcome and lower adverse effect than steroid injection.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blinded controlled study. Patients with the diagnosis of trigger finger will be recruited and enrolled from Taipei Veteran General Hospital PM&R outpatient clinic. Subjects will be randomized into two groups; hyaluronic acid and triamcinolone acetonide injections, both via ultrasound-guided with one injection only.We hypothesize that through the anti-inflammatory property of the hyaluronate acid, the treatment effects will be as effective as the traditionally used steroid injections with equal or even lower recurrence rate for treatment of trigger finger. We expect that injections of hyaluronate into tendon sheath could become a new treatment option for trigger finger.

ELIGIBILITY:
Inclusion Criteria:

* patients with trigger digits and patients
* without previous treatment of the trigger digit

Exclusion Criteria:

* patients with prior treatment of the trigger digit (eg, splinting, injection, or therapy),
* patients less than
* 20 years old,
* patients with allergy or contraindication to hyaluronic acid,
* patients with trigger digits due to rheumatoid arthritis,
* and patients with infection at the site of injection.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Quinnell classification | Pre-injection; 3-weeks and 3-months post-injections
  he Quinnell system grades trigger fingers as:
  0 - normal movement
  1. - uneven movement
  2. - locking can be corrected with active motion
  3. - locking corrected with passive motion
  4. - unable to correct deformity

SECONDARY OUTCOMES:
hand functional evaluation | Pre-injection; 3-weeks and 3-months post-injections
  using the Michigan Hand Outcome Questionnaire (MHQ)
visual analog scale | Pre-injection; 3-weeks and 3-months post-injections
total active motion (TAM) | Pre-injection; 3-weeks and 3-months post-injections
  Deﬁ ned as the total ROM achieved when all three joints-metacarpophalangeal (MCP), proximal interphalangeal (PIP) and distal interphalangeal (DIP) of a digit are actively ﬂ exed or extended simultaneously, minus any extension deﬁ cit at any of the three joints
grip strength | Pre-injection; 3-weeks and 3-months post-injections
  dynamometer strength test (JAMAR grip)

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Lan Kao, MD, PhD, Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Liu DH, Tsai MW, Lin SH, Chou CL, Chiu JW, Chiang CC, Kao CL. Ultrasound-Guided Hyaluronic Acid Injections for Trigger Finger: A Double-Blinded, Randomized Controlled Trial. Arch Phys Med Rehabil. 2015 Dec;96(12):2120-7. doi: 10.1016/j.apmr.2015.08.421. Epub 2015 Sep 1. PMID 26340807